CLINICAL TRIAL: NCT04119206
Title: Comparison of the Vasopressin-2 Antagonist Tolvaptan and Fluid Restriction in the Treatment of Hyponatremia Following Pituitary Surgery
Brief Title: Tolvaptan Versus Fluid Restriction in SIADH
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Andrea Kleindienst, MD, PhD, Associate Professor, University of Erlangen-Nürnberg Medical School
Other Study IDs: Tolvaptan
Record Dates: First submitted 2019-10-02; First posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Hyponatremia; Syndrome of Inappropriate ADH (SIADH) Secretion; Pituitary
Keywords: hyponatremia; vasopressin; anti-diuretic hormone; fluid restriction; tolvaptan; pituitary surgery
MeSH Terms: conditions — Hyponatremia; Inappropriate ADH Syndrome; Pituitary Diseases; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: Normonatremic control, no intervention.
- Fluid restriction: Hyponatremic patients (serum sodium <135mmol/L): restriction of fluid intake < 1L
- Tolvaptan 3.75mg: Hyponatremic patients (serum sodium <135mmol/L): tolvaptan 3.75 mg tablet; The serum sodium concentration was controlled at 6:00 pm. Those patients, whose serum sodium concentration further dropped below 132 mmol/L, were treated with a second tablet of tolvaptan and the serum sodium was measured the next day at 8:00 am. Those patients, whose serum sodium was increased by not more than 5 mmol/L underwent the next blood check on the next day at 8:00 am. Those patients, whose serum sodium increased by more than 5 mmol/L were treated by 1L tea/water or a 500 mL 5% glucose infusion.
- Tolvaptan 7.5mg: Hyponatremic patients (serum sodium <135mmol/L): tolvaptan 7.5 mg tablet; The serum sodium concentration was controlled at 6:00 pm. Those patients, whose serum sodium concentration further dropped below 132 mmol/L, were treated with a second tablet of tolvaptan and the serum sodium was measured the next day at 8:00 am. Those patients, whose serum sodium was increased by not more than 5 mmol/L underwent the next blood check on the next day at 8:00 am. Those patients, whose serum sodium increased by more than 5 mmol/L were treated by 1L tea/water or a 500 mL 5% glucose infusion.

SUMMARY:
Context. The relevance of hyponatremia has been acknowledged by guidelines from the United States of America (2013) and Europe (2014). However, treatment recommendations differ due to limited evidence.

Objective. In hyponatremia following pituitary surgery - caused by the syndrome of inappropriate antidiuretic hormone (SIADH) secretion - the investigators compared fluid restriction with the pharmacological increase of water excretion by blocking the vasopressin 2 receptors with tolvaptan at a low and moderate dose.

Design. Prospective observational study.

Setting. Neurosurgical Department of a University hospital with more 200 pituitary procedures per year.

Patients. Participants undergoing surgery for sellar lesions and developing a serum sodium below 135 mmol/L. The diagnosis of SIADH was established by eu- or hypervolemia (daily measurement of body weight and fluid balance daily), an inappropriately concentrated urine (specific gravity) and exclusion of a cortico- and thyreotropic insufficiency.

Intervention. Participants were treated with fluid restriction (n=38) or tolvaptan at 3.75 (n=38) or 7.5 mg (n=48) orally.

Main Outcome Measures. Treatment efficacy was assessed by the duration of hyponatremia, sodium nadir and length of hospitalization. Safety was established by an increment serum sodium below 10 mmol/L per day and exclusion of side effects.

DETAILED DESCRIPTION:
Patients of the Department of Neurosurgery, University of Erlangen-Nuremberg, undergoing surgery for sellar lesions were prospectively included. The study protocol was approved by the local Ethical Committee (Re.-No. 103_12 BC). Informed written consent was given by the participants or the next-of-kin in each case. Exclusion criteria comprised of those below 18 years of age, pregnancy and a drug intolerance.

Patients Baseline information included age, gender, BMI and the clinical presentation. The pre-operative work-up included an opthalmological examination, a 1.5 Tesla magnetic resonance imaging (MRI) with 2mm axial, coronal and sagittal sections revealing the tumor localization, extension, and its invasive behavior. Microsurgery was always performed by the same surgeon. The macroscopic delineation and invasiveness, the surgical manipulation of the pituitary stalk and extend of tumor resection, surgical complications, as well as an intraoperative cerebrospinal fluid (CSF) leak were documented. The tumor and the dura of the floor of the sella were examined histo-pathologically including the proliferation rate, regressive changes, atypical findings, and the existence of Crooke cells and periodic acid-Schiff (PAS) expression. Routine laboratory work-up included creatinine, urea, and alanine aminotransferase (ALT).

The pre- and postoperative endocrine testing of the pituitary function comprised the basal values of cortisol (CORT), growth hormone (GH), insulin-like growth factor (IGF) 1, thyroid stimulating hormone (TSH), free thyroxine (fT4), total triiodothyronine (tT3), luteinizing hormone (LH), follicle stimulating hormone (FSH), testosterone (TES), estradiol (E2), and prolactin (PRL). Insufficiency of the corticotropic axis was determined by a short synacthen test (adreno-corticotropic hormone; ACTH)-test stimulating with 0.25 mg Syntropin (Synacthen, Novartis Pharma, Nuremberg, Germany) intra-venously and serum cortisol measurement at 0 and 30 minutes.

Surveillance Post-operatively, participants were transferred to the general floor. For a minimum of 10 days, fluid intake, body weight, and urine volume with specific gravidity are documented daily, along with blood pressure and heart rate three-times daily, blood samples for the assessment of electrolytes are taken on day 1, 2, 3, 5, 7, and 9. An endocrine dynamic testing was performed on day 7.

Analytical methods Venous blood samples were drawn in the morning between 7:00 and 9:00 am into pre-cooled tubes. Clotted samples were promptly centrifuged at 3,000 X g for 15 min at 4 degree Celsius, and then the plasma was frozen at -80 degree Celsius until analysis.

An automated system (Immulite®2000, Diagnostic Products Corporation) was used for the following serum hormone measurements: Serum cortisol levels > 10.5 µg/dL, with an assay sensitivity of 0.20 µg/dL, was considered normal; a cortisol response peak to the ACTH-test higher than 18 µg/dl was considered adequate; for IGF-1 of 135-485 ng/mL (18-30 years), 120-397 ng/mL (31-40 years), 113-306 ng/mL (41-50 years), 100-250 ng/mL (51-60 years), and 92-229 ng/mL (>60 years) (assay sensitivity of 20 ng/mL); LH > 0.25 U/L (follicular phase) and > 20 U/L (menopausal) in women, and > 1 international units (IU)/L in men (assay sensitivity of 0.05 mIU/mL); FSH > 0.25 U/L (follicular phase) and > 30 U/L (menopausal) in women, and > 1 IU/L in men (assay sensitivity of 0.1 mIU/mL); TES > 90 ng/dL in men (assay sensitivity of 15 ng/dL); E2 > 60 pg/mL (follicular phase) and > 10 pg/mL (menopausal) in women (assay sensitivity of 15 pg/mL); PRL < 500 micro international units (µIU)/L (assay sensitivity of 0.16 µU/L); PRL serum concentrations were considered normal < 360 ng/ml in men and < 530 ng/mL in women. TSH serum concentrations were considered normal > 0.45 µU/mL, fT4 > 0.77 ng/dL, and tT3 > 0.8 ng/mL.

Study design Treatment of hyponatremia was initiated as soon as a SIADH was confirmed by eu- or hypervolemia (daily measurement of body weight and fluid balance), an inappropriately concentrated urine (measurement of specific gravity), and exclusion of a cortico- and thyreotropic insufficiency. The established treatment regime consisted of a restriction of fluid intake < 1 L whenever the serum sodium dropped below 135 mmol/L or the body weight gained more than 1 kg (fluid restriction). In a second cohort of patients, the fluid restriction was replaced by a low dosage of tolvaptan (tolvaptan 3.75 mg), and in a third cohort by a medium dosage (tolvaptan 7.5 mg). Since a rapid correction of hyponatremia is hazardous and leaves the patient vulnerable to the risk of osmotic demyelination, we not only started the cohort study with a very low concentration of 3.75 mg tolvaptan, but also established a tight follow-up regime after medication. The serum sodium concentration was controlled at 6:00 pm. Those participants, whose serum sodium concentration further dropped below 132 mmol/L, were treated with a second tablet of tolvaptan and the serum sodium was measured the next day at 8:00 am. Those participants, whose serum sodium was increased by not more than 5 mmol/L underwent the next blood check on the next day at 8:00 am. Those participants, whose serum sodium increased by more than 5 mmol/L were treated by 1L tea/water or a 500 mL 5% glucose infusion.

Statistical analysis SPSS statistical software (SPSS Inc., Chicago, Illinois, USA) was used for all statistical analyses. Analyses were performed using the Chi-squared test and Mann-Whitney U tests where appropriate. Significance was accepted at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

Informed written consent was given by the participant or the next-of-kin.

Exclusion Criteria:

Age below 18 years Pregnancy Tolvaptan intolerance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Department of Neurosurgery, University of Erlangen-Nuremberg, undergoing surgery for sellar lesions were prospectively included.
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Mean serum sodium concentration | Day 1 post-op up to 15 days
  Postoperative mean serum sodium
Serum sodium nadir concentration | Day 1 post-op up to 15 days
  Postoperative serum sodium nadir
Number of days with serum sodium concentration below 136mmol/L | Day 1 post-op up to 15 days
  No. of postoperative days serum sodium was below 136mmol/L
Number of days with serum sodium concentration below 133mmol/L | Day 1 post-op up to 15 days
  No. of postoperative days serum sodium was below 133mmol/L

SECONDARY OUTCOMES:
Number of events with mild serum sodium overcorrection | Day 1 post-op up to 15 days
  Serum sodium overcorrection > 5mmol/L*24hrs
Number of events with severe serum sodium overcorrection | Day 1 post-op up to 15 days
  Serum sodium overcorrection > 10mmol/L*24hrs
Number of days in the hospital | Up to 1 month
  Duration of hospital stay